CLINICAL TRIAL: NCT05510895
Title: Neoadjuvant Encorafenib, Binimetinib and Cetuximab for Patients With BRAF V600E Mutated/pMMR Localized Colorectal Cancer
Acronym: NeoBRAF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Pierre Fabre Pharma GmbH (Industry); Merck Serono GmbH, Germany (Industry); Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIO-KRK-0420
Record Dates: First submitted 2022-08-17; First posted 2022-08-22 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer; Colon Cancer; BRAF V600E; BRAF V600 Mutation; Localized Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — binimetinib; encorafenib; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neoadjuvant and adjuvant triplet combination of encorafenib, binimetinib and cetuximab (Experimental): Neoadjuvant treatment with encorafenib, binimetinib and cetuximab for up to 8 weeks (4 biweekly cycles). In Week 10-12 surgery of the tumor followed by central determination of tumor regression grade (TRG).
  TRG0-1: insufficient response to neoadjuvant triplet. Standard chemotherapy with fluoropyrimidines and oxaliplatin should be applied. TRG2-4: 4-8 weeks after surgery adjuvant treatment with encorafenib, binimetinib and cetuximab continues for up to 16 Weeks (8 biweekly cycles).
  Interventions: Drug: Binimetinib

INTERVENTIONS:
Drug: Binimetinib — Triplet combination administered neoadjuvant and adjuvant, depending on TRG
  Other Names: Encorafenib; Cetuximab

SUMMARY:
AIO-KRK-0420 NeoBRAF is a single arm, multicenter, phase II trial with neoadjuvant encorafenib, binimetinib and cetuximab for patients with BRAF V600E mutated/pMMR localized colorectal cancer.

DETAILED DESCRIPTION:
This is a single arm, multicenter, phase II trial for patients with unresected BRAF V600E mutated/pMMR localized colorectal cancer (CRC). Patients enrolled will be treated with neoadjuvant encorafenib (300mg QD), binimetinib (45mg BID) and cetuximab (500mg/m² biweekly) for 8 weeks. Neoadjuvant treatment will be followed by surgery. First Endpoint is TRG (Tumor-Regression-Grade) which will be analyzed centrally. Patients with TRG>1 will receive adjuvant treatment with encorafenib (300mg QD), binimetinib (45mg BID) and cetuximab (500mg/m² biweekly) for up to 16 weeks. For patients with TRG<2 EOT will be reached 4-6 weeks after last dosage of encorafenib, binimetinib and cetuximab and further treatment is at investigator discretion (CAPOX recommended). All subjects will be followed every 3 months after surgery for up to 4 years after start of recruitment.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-confirmed adenocarcinoma of the colon or upper rectum if too high for radiotherapy.
2. Radiologically (CT/MRI) staged disease as: T3-4 (as invasion of surrounding tissue structures or organs) and/or nodal positive (N+ defined as regional lymph node(s) without fat hilus and short axis diameter of ≥1 cm), M0.
3. BRAF V600E mutation and pMMR or MSS (as determined by a validated test, preferably PCR or NGS).
4. ECOG performance status ≤ 1.
5. Age ≥ 18 years.
6. Adequate hematologic function at screening as follows:

   ANC ≥ 1.5 x 109/L, platelets ≥ 100 x109/L, hemoglobin ≥ 9.0 g/dL.
7. Adequate liver function at screening as measured by serum transaminases (AST & ALT) ≤ 2.5 x ULN and total bilirubin ≤ 1.5 x ULN. Patients with known Gilbert disease who have serum bilirubin level ≤ 3 × ULN may be enrolled.
8. Adequate renal function at screening: serum creatinine ≤ 1.5 x ULN.
9. Adequate serum electrolytes at screening defined as serum potassium and magnesium levels within institutional normal limits (Note: replacement treatment to achieve adequate electrolytes will be allowed.
10. Adequate cardiac function at screening characterized by left ventricular ejection fraction (LVEF) ≥ 50% as determined by ECHO and QT interval corrected for heart rate using Fridericia's formula (QTcF) value ≤ 480 msec.
11. Negative serum pregnancy test at screening for women of childbearing potential.
12. Highly effective contraception for both male and female subjects if the risk of conception exists. (Note: The effects of the trial drugs on the developing human fetus are unknown; thus, women of childbearing potential and men able to father a child must agree to use highly effective contraception, defined as methods with a failure rate of less than 1 % per year, containing at least 1 form of non-hormonal contraception. Highly effective contraception is required at least 28 days prior, throughout and for at least 6 months after interventional study treatment (encorafenib, binimetinib and cetuximab).
13. Signed and dated written informed consent.
14. Ability to take oral medication.
15. Ability to comply with the protocol for the duration of the study, including hospital/office visits for treatment and scheduled follow-up visits and examinations.

Exclusion Criteria:

1. Any prior systemic therapy, surgery or radiotherapy of the colorectal cancer disease.
2. History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO (e.g., uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes).
3. Malignancies other than disease under study within 5 years prior to inclusion, with the exception of those with a negligible risk of metastasis or death (e.g., expected 5-year OS >90%) treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, localized prostate cancer treated surgically with curative intent, ductal carcinoma in situ treated surgically with curative intent).
4. Known severe hypersensitivity reactions to monoclonal antibodies or BRAF-/MEK-inhibitors (grade ≥ 3 NCI-CTCAE v 5), any history of anaphylaxis, or uncontrolled asthma (that is, 3 or more features of partially controlled asthma).
5. Pregnancy or lactation.
6. Known alcohol or drug abuse.
7. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (≤ 6 months prior to enrolment); myocardial infarction (≤ 6 months prior to enrolment), acute coronary syndromes [including unstable angina, coronary artery bypass graft (CABG), coronary angioplasty or stenting) ≤ 6 months prior to enrolment]; congestive heart failure (≥New York Heart Association Classification Class II); or history or current evidence of clinically significant arrhythmia and/or conduction abnormality (≤ 6 months prior to enrolment), except rate controlled atrial fibrillation and paroxysmal supraventricular tachycardia.
8. Uncontrolled hypertension defined as persistent elevation of systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg despite current therapy.
9. Preexisting interstitial lung disease.
10. Impaired GI function or disease that may significantly alter the absorption of encorafenib or binimetinib (e.g., ulcerative diseases, uncontrolled vomiting, malabsorption syndrome, small bowel resection with decreased intestinal absorption).
11. History of thromboembolic or cerebrovascular events ≤ 6 months prior to enrolment, including transient ischemic attacks, cerebrovascular accidents, deep vein thrombosis or pulmonary emboli.
12. Concurrent neuromuscular disorder that is associated with the potential of elevated CK (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy).
13. Known human immunodeficiency virus (HIV) infection or active hepatitis B or C infection.
14. All other significant diseases, which, in the opinion of the Investigator, might impair the subject's tolerance of trial treatment.
15. Any psychiatric condition that would prohibit the understanding or rendering of informed consent.
16. Any approved anticancer therapy, including chemotherapy, hormonal therapy or radiotherapy, within 5 half-lives or 4 weeks (the longer period applies) prior to initiation of study treatment.
17. Current treatment with a non-topical medication or current intake of herbal preparations / supplements / foods known to be a strong inhibitor of CYP3A4. However, patients who either discontinue such treatment/intake or switch to another medication at least 7 days prior to starting study treatment are eligible.
18. Concomitant use of St. John's Wort (hypericum perforatum).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Tumor regression grade (TRG) | immediately after the surgery
  Tumor regression will be centrally graded according to the grading system developed by Dworak et al (Dworak, Keilholz et al. 1997).

SECONDARY OUTCOMES:
Safety and tolerability (acc. to NCI CTC AE v5.0) incl. vital signs, clinical parameters and overall feasibility of the regimen | max 54 months
  Safety assessments will include physical examinations including visual and skin assessment as well as vital signs (blood pressure, heart rate, respiratory rate), performance status (ECOG), clinical laboratory profile, 12-lead ECG and ECHO, ophthalmologic assessment, concomitant medication/therapies/procedures and adverse events. All observed adverse events will be graded according to NCI CTCAE v5. Adverse events will be analysed overall and concerning their potential relationship to study treatment and surgical intervention. Serious adverse events (SAE) will be analysed in the same way.
Perioperative morbidity and mortality | max 24 months
  Perioperative morbidity and mortality are defined as prolongation of hospitalization (discharge >20 days after surgery), re-hospitalization or reoperation under general anaesthesia within 30 days of surgery or death during surgery or within 30 days of surgery; Other severe postoperative complications within 30 days of surgery including surgery-associated bleeding with replacement ≥ 4 units of erythrocyte concentrates, transient liver failure, defined as a bilirubin level >10 mg/dL lasting > 7 days, renal failure requiring dialysis, respiratory failure with renewed necessary mechanical ventilation or >26 h, necessary mechanical ventilation, deep venous thromboembolism, cardiac failure, major impaired wound healing necessitating re-operation or prolonging hospitalization (discharge >20 days after surgery); >8 weeks delay of surgery due to study treatment-related toxicity; and further.
R0-resection rate | max 24 months
  The R0 resection rate will be determined as the rate of R0 resections out of all resected patients. In addition, the R1 and/or R2 resection rates will be determined.
Overall Response Rate (ORR) according to RECIST v1.1 | max 54 months
  Response rate to preoperative treatment will be assessed according to RECIST v1.1.
Disease free survival | max 54 months
  Disease free survival will be determined as time from start of study treatment to date of first observed disease recurrence (either local or distant) or death from any cause.
Overall survival (OS) | max 54 months
  Overall survival will be determined as time from start of study treatment to date of death from any cause.
Translational research 1 | max 54 months
  Correlation of quantitative BRAF V600E levels (measured by ddPCR) with TRG
Translational research 2 | max 54 months
  Evaluation of mechanism of relative resistance in patients with less response (evaluated by tumor and liquid biopsy NGS profiling at baseline and after treatment)
Translational research 3 | max 54 months
  Comparison of ctDNA clearance and TRG with a BRAF mutant/pMMR cohort from the planned neoadjuvant PROTECTOR study receiving neoadjuvant chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Stein, Prof. Dr., Principal Investigator — Hämatologisch-Onkologische Praxis Eppendorf, 20249 Hamburg, Germany
Locations (1):
- Hämatologisch-Onkologische Praxis Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Working Group for Medical Oncology from the German Cancer Society — https://www.aio-portal.de/
- See also: AIO-Studien-gGmbH — https://www.aio-studien-ggmbh.de/